CLINICAL TRIAL: NCT00845364
Title: Metabolic Support With Perhexiline to Protect Myocardium Undergoing Coronary Artery Surgery
Acronym: CASPER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Birmingham (Other)
Collaborators: University of Birmingham (Other); Brighton and Sussex University Hospitals NHS Trust (Other); British Heart Foundation (Other)
Responsible Party: Mr Domenico Pagano, University Hospital Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RRK3217; Eudract 2006-003164-62; REC 06/Q0104/141; BHF PG/06/044/20703
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: Myocardial Reperfusion Injury; Cardiac Output, Low
Keywords: Perhexiline; Coronary artery bypass; Myocardial reperfusion injury; Cardiac output, low; Troponin
MeSH Terms: conditions — Myocardial Reperfusion Injury; Cardiac Output, Low | interventions — Perhexiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perhexiline (Experimental): Pre-operative administration of Perhexiline tablets according to dosing schedule
  Interventions: Drug: Perhexiline
- Placebo (Placebo Comparator): Pre-operative administration of placebo tablets according to dosing schedule
  Interventions: Drug: Placebo marked PEXSIG

INTERVENTIONS:
Drug: Perhexiline — Tablets. Dose: 200mg BD for 3 days, then 100mg BD until surgery. Duration of therapy: 5-31 days.
  Other Names: PEXSIG
  Arms: Perhexiline
Drug: Placebo marked PEXSIG — Tablets. Dose: 200mg BD for 3 days, then 100mg BD until surgery. Duration of therapy: 5-31 days.
  Arms: Placebo

SUMMARY:
Open-heart surgery causes injury of the heart muscle. Although this is usually mild, temporary and reversible, if it is severe it can endanger life and require additional high cost care. During surgery, techniques are used to protect the heart from injury, but these remain imperfect. This study assesses the effect of facilitating sugar metabolism (a more efficient fuel) by the heart muscle using the drug Perhexiline given before the operation. This treatment has a sound experimental basis for improving outcome. If this improvement is confirmed surgical results could be improved. The investigators will be studying heart function, heart muscle energy stores and chemicals which quantify the amount of heart muscle injury. The investigators' hypothesis is that Perhexiline will improve the protection of the heart by decreasing damage that may occur during heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* First-time
* Isolated coronary artery bypass surgery

Exclusion Criteria:

* Diabetes Mellitus
* Renal impairment with Creatinine greater than or equal to 200micromol/L
* Atrial fibrillation
* Amiodarone therapy, recent (in last month) or current
* Hepatic impairment, significant preoperative
* Peripheral neuropathy
* Pregnancy or breast-feeding
* Emergency surgery or required on clinical grounds within 5 days of referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2007-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Low Cardiac Output Syndrome | 6 hours post-removal of aortic X-clamp

SECONDARY OUTCOMES:
Increase in Cardiac index of greater than or equal to 0.3 L/min/m2 | 6 hours post-removal of aortic X-clamp
Incidence of inotropes use according to protocol | 6 and 12 hours post-removal of aortic X-clamp
Peak and total release of Troponin | 6, 12 and 24 hours post-release of aortic X-clamp

CONTACTS AND LOCATIONS:
Overall Officials: Domeinco Pagano, MD FRCS, Principal Investigator — University Hospital Birmingham
Locations (2):
- United Kingdom (2):
  - University Hospital Birmingham, Birmingham, West Midlands
  - Brighton & Sussex University Hospitals NHS Trust, Brighton, West Sussex

REFERENCES:
- [Background] Quinn DW, Pagano D, Bonser RS, Rooney SJ, Graham TR, Wilson IC, Keogh BE, Townend JN, Lewis ME, Nightingale P; Study Investigators. Improved myocardial protection during coronary artery surgery with glucose-insulin-potassium: a randomized controlled trial. J Thorac Cardiovasc Surg. 2006 Jan;131(1):34-42. doi: 10.1016/j.jtcvs.2005.05.057. PMID 16399292
- [Background] Ranasinghe AM, Quinn DW, Pagano D, Edwards N, Faroqui M, Graham TR, Keogh BE, Mascaro J, Riddington DW, Rooney SJ, Townend JN, Wilson IC, Bonser RS. Glucose-insulin-potassium and tri-iodothyronine individually improve hemodynamic performance and are associated with reduced troponin I release after on-pump coronary artery bypass grafting. Circulation. 2006 Jul 4;114(1 Suppl):I245-50. doi: 10.1161/CIRCULATIONAHA.105.000786. PMID 16820580
- [Background] Ashrafian H, Horowitz JD, Frenneaux MP. Perhexiline. Cardiovasc Drug Rev. 2007 Spring;25(1):76-97. doi: 10.1111/j.1527-3466.2007.00006.x. PMID 17445089
- [Derived] Drury NE, Howell NJ, Calvert MJ, Weber RJ, Senanayake EL, Lewis ME, Hyde JA, Green DH, Mascaro JG, Wilson IC, Graham TR, Rooney SJ, Viant MR, Freemantle N, Frenneaux MP, Pagano D; investigators. The effect of perhexiline on myocardial protection during coronary artery surgery: a two-centre, randomized, double-blind, placebo-controlled trial. Eur J Cardiothorac Surg. 2015 Mar;47(3):464-72. doi: 10.1093/ejcts/ezu238. Epub 2014 Jun 19. PMID 24948413